CLINICAL TRIAL: NCT04604743
Title: Exploratory Sequential Mixed Methods Cluster Randomized Controlled Implementation Science Trial to Develop a Clinic-based HPV and COVID-19 Vaccine Promoting Intervention for African American Older Adolescents in Rural Alabama
Brief Title: Clinic-based HPV and COVID-19 Vaccine Promoting Intervention for AfAm Adolescents in Alabama
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: PI transferred institutions; the grant was not transferred to the new university.
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Henna Budhwani, Assistant Professor, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: MISP #60590
Record Dates: First submitted 2020-10-25; First posted 2020-10-27 (Actual); Last update posted 2023-04-06 (Actual); Status verified 2023-04

CONDITIONS: Vaccine Refusal
MeSH Terms: conditions — Vaccination Refusal | interventions — Methods

STUDY DESIGN:
Intervention Model Description: 2) Cluster randomized controlled trial design (N=4 clinics). This design minimizes risk of contamination between participants in different arms and is ideal when settings are similar in population characteristics. Cluster randomized controlled trials are frequently used when interventions are to be carried out at the level of whole groups (clinic populations).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): 2 Clinics
  Interventions: Behavioral: Intervention, TBN
- Control (No Intervention): 2 Clinics

INTERVENTIONS:
Behavioral: Intervention, TBN — The intervention will target adolescents aged 15-17 years who have not received at least one dose of the HPV vaccine. The intervention has yet to be named; this will occur through the conduct of Aim 1. Our intervention, when developed, will improve knowledge of HPV, COVID-19, the HPV vaccine, and the COVID-19 vaccine (Information), reduce stigma and distrust improving motivation (Motivation), leading to improved vaccine confidence and higher vaccination rates and lower vaccine hesitancy (Behavioral Skills). Each one of these three change objectives will be encapsulated in its own Zoom-based session with the near peer interventionist. We anticipate that each modular session will be no longer than seven minutes; thus, the entire three module intervention will be no longer than twenty-one minutes long.
  Arms: Intervention

SUMMARY:
In this 30-month study, the investigators propose to develop a culturally appropriate vaccine confidence intervention, targeting positive change related to HPV vaccine uptake behavior and reducing sentiments of hesitancy towards a COVID-19 vaccine, that can be seamlessly integrated into the existing environment of pediatric and family practice clinics in rural Alabama. To do so, the investigators will first assess stakeholders' knowledge, sentiments, and beliefs related to vaccination in general, a COVID-19 vaccination, and the HPV vaccination. The investigators will also assess stakeholders' perceptions of barriers to vaccination that exist in rural Alabama. This will occur in Aim 1. Then, in Aim 2, the investigators will use these data to inform the development of a non-invasive, modular synchronous counseling intervention targeting 15-17 year old adolescents (rationale for this age range presented later in this proposal). After the intervention has been finalized, in our final aim, Aim 3, we will conduct a hybrid type 1 effectiveness-implementation cluster randomized control trial to assess intervention acceptability and feasibility (N=4 clinics; N=120 adolescents), while also assessing for a "clinical signal" of effectiveness. To support dissemination and scale up, also during Aim 3, we will document implementation contexts to provide real-world insight. To do this, the investigators will conduct in-depth interviews with the same groups of stakeholders that we interviewed in Aim 1.

DETAILED DESCRIPTION:
In this 30-month study, the investigators propose to develop a culturally appropriate vaccine confidence intervention, targeting positive change related to HPV vaccine uptake behavior and reducing sentiments of hesitancy towards a COVID-19 vaccine, that can be seamlessly integrated into the existing environment of pediatric and family practice clinics in rural Alabama. To do so, the investigators will first assess stakeholders' knowledge, sentiments, and beliefs related to vaccination in general, a COVID-19 vaccination, and the HPV vaccination. The investigators will also assess stakeholders' perceptions of barriers to vaccination that exist in rural Alabama. This will occur in Aim 1. Then, in Aim 2, the investigators will use these data to inform the development of a non-invasive, modular synchronous counseling intervention targeting 15-17 year old adolescents (rationale for this age range presented later in this proposal). After the intervention has been finalized, in our final aim, Aim 3, we will conduct a hybrid type 1 effectiveness-implementation cluster randomized control trial to assess intervention acceptability and feasibility (N=4 clinics; N=120 adolescents), while also assessing for a "clinical signal" of effectiveness. To support dissemination and scale up, also during Aim 3, we will document implementation contexts to provide real-world insight. To do this, the investigators will conduct in-depth interviews with the same groups of stakeholders that we interviewed in Aim 1.

ELIGIBILITY:
Inclusion Criteria:

* Ages 15-26 years
* Have not completed HPV vaccination schedule
* Located in a rural, non-urban setting
* Able to provide informed consent

Exclusion Criteria:

* Doe not meet inclusion criteria

Ages: 15 Years to 26 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 0 (Actual)
Dates: Start 2021-04-20 (Actual); Primary Completion 2022-08-07 (Actual); Study Completion 2022-08-07 (Actual)

PRIMARY OUTCOMES:
HPV Vaccination | Within 6 months from intervention
  Initial dose of HPV vaccine within 6 months from intervention
Reduction in Vaccine Hesitancy | Within 6 months from intervention
  Reduction in hesitancy measured by change in knowledge and motivation via surveys; survey tools to be developed based on qualitative data

CONTACTS AND LOCATIONS:
Locations (1):
- University of Alabama at Birmingham (UAB), Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: No
Data sharing with occur in compliance with Merck's data sharing policy.

REFERENCES:
- [Derived] Budhwani H, Sharma V, Long D, Simpson T. Developing a Clinic-Based, Vaccine-Promoting Intervention for African American Youth in Rural Alabama: Protocol for a Pilot Cluster-Randomized Controlled Implementation Science Trial. JMIR Res Protoc. 2022 Apr 8;11(4):e33982. doi: 10.2196/33982. PMID 35212640